CLINICAL TRIAL: NCT01424605
Title: The Comparison of Glidescope® and the Direct Laryngoscopy in the Insertion of the Double Lumen Endotracheal Tube
Acronym: Glidescope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hung-Te Hsu (980393), visiting stuff , department of anesthesia, Kaohsiung Medical University Chung-Ho Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KMUH-IRB-980393; KMUH-IRB-980393 (Other: KaohsiungMU)
Record Dates: First submitted 2011-05-18; First posted 2011-08-29 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Anesthesia Intubation Complication
Keywords: left-sided double lumen bronchial tube; GlideScope videolaryngoscope; direct laryngoscope
MeSH Terms: interventions — Intubation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DLT intubation (Experimental)
  Interventions: Procedure: DLT intubation

INTERVENTIONS:
Procedure: DLT intubation — Using a video-assisted laryngoscope to facilitate endotracheal tube intubation
  Other Names: Intubation with GlideScope

SUMMARY:
Double-lumen bronchial tube (DLT) had been demonstrated to benefit for thoracic surgery and also played an important role to achieve one-lung ventilation (OLV) for exploring the surgical fields. However, compared with the single-lumen endotracheal tube (SLT), the DLT had larger OD (outer diameter), longer length, and was more complex in its structure. For avoiding oral tissue trauma and shortening the DLT intubating time, thus, an adequate and complete glottic viewing under laryngoscope was needed.

Over the past decade, several video-assisted laryngoscopes had been developed to facilitate the tracheal intubation in the difficult airway. Among these devices, the GlideScope® videolaryngoscope (GVL) (Verathon, Bothell, WA, USA) was a reusable video laryngoscope with a 60° curvature blade. A light source and a digital video camera were installed at the tip of the laryngoscope blade and the pictures of the glottis and the vocal cords were displayed on an LCD monitor. We could insert the endotracheal tube passing the vocal cords into the trachea more precisely and had less tissue damaging under the GVL's guidance.

Compared with direct MacIntosh laryngoscope, the GVL had been reported that it can decrease the intubation time and increase the successful rate of first intubation in normal and difficult airways. However, the efficacy of the GVL in intubating the DLT was unclear and had never been evaluated. Therefore, the aim of this study was to compare the intubation conditions, safety, and patient comfort between using the GVL and the direct Macintosh laryngoscope in a specific population of patients needed DLT intubation. Main outcome measures were intubation success rates and the time needed to intubate the DLT with the two devices.

DETAILED DESCRIPTION:
The study protocol was approved by the Institutional Research Board of the Memorial Hospitals of Kaohsiung Medical University and all patients included in the study gave written informed consent. Sixty patients with American Society of Anesthesiologists physical status I-III, ≧ 18 years of age, and needed double-lumen endotracheal tube (DLT) for thoracic surgery were enrolled in this study. Exclusion criteria were increased risk for regurgitation and pulmonary aspiration, history of gastroesophageal reflux, and pregnancy. Furthermore, when a tracheostomy or prolonged ventilation on ICU was planned, patients were also excluded. All tracheal intubations in the study were performed by two experienced (> 10 year) Board Certified anesthesiologists who each had experience of at least 300 tracheal intubations with each device before starting the study.

After the patient had entered the operating room, standard monitoring including ECG, invasive blood pressure measurement on the radial artery and pulse oximetry were established. Patients were randomly assigned to direct MacIntosh laryngoscope group (Group M, n = 30) or GVL group (Group G, n = 30) by opening a sealed envelope after they had entered the operating theatre. Anesthesia was induced with propofol 2-3 mg.kg-1, fentanyl 2μg.kg-1, and rocuronium 0.6mg.Kg-1. After achieving adequate muscle relaxation and anesthetic depth, DLT intubation was performed with direct laryngoscope or GVL. The bronchial and the tracheal cuff of the DLT were lubricated with SURGILUBE® sterile, surgical lubricant (E. FOUGERA & CO. Melville, New York, A division of Nycomed US Inc.) thinly before intubation.

Measurements The demographic characteristics of both groups included age (years), gender (female/male), weight (kg), height (cm), body mass index (BMI), and ASA classification were recorded. The airway characteristics included the modified Mallampati classification, mouth opening (active and passive), and the thyromental distance were also recorded. Patients were measured of thyromental distance and incisor gap on maximal opening of the mouth and grading of The modified Mallampati classification in the operative room by another anesthesiologist not involved in the study. Passive mouth opening was measured after induction of anesthesia. After pre-oxygenation with oxygen 100%, patients received thiamylal 5 mg.kg-1 and fentanyl 2μg.kg-1 for anesthesia induction and facilitated DLT intubation with rocuronium 0.8 mg.kg-1 and propofol 1.0 mg.kg-1.

The total time to calculate DLT insertion (T3) was separated into T1 and T2, respectively, defined as started after jaw opening when the GVL or the direct laryngoscope passed the patient's lips and stopped when three complete waves of end-tidal CO2 showed on the monitor of capnography and measured by an independent observer. T1 time interval was calculated from the jaw opening, placement of GVL or standard Macintosh laryngoscope, to the view of glottis opening. T2 time interval was calculated from intubator holding DLT to three complete waves of end-tidal CO2 showed on the monitor of capnography. The procedures to position of DLT were declared in brief as following: the distal 10-12cm of the DLT was curved to approximately 90°; a conventional laryngoscope in group M and a Glidescope in group G to assist position DLT into trachea [4]; the tip of the DLT bronchial lumen was passed through the vocal cords and advanced into the glottis; to remove stylet of DLT; 180° counterclockwise rotation to facilitate the insertion of the bronchial cuff and tracheal lumen past the vocal cords; an additional 90° clockwise rotation to fit the tube into left main bronchus [5]. Grading of laryngo-pharyngeal tissues viewed by intubator according to the Cormack and Lehane classification (grades I-IV) that defined as grade I- complete glottis visible, grade II- anterior glottis not seen, grade III- epiglottis seen, but not glottis, and grade IV- epiglottis not seen [6]. The intubator determined the grades of laryngeal viewing either by direct laryngoscope or by Glidescope® with video monitor. The backwards upwards rightwards pressure (BURP) maneuver to optimize the glottis view was also recorded and the pressure grading was defined as none, light, and heavy.

After the blade of laryngoscope or GlideScope® was removed, we examined blood coating on its surface. The oral cavity, pharynx and larynx for signs of lacerations or bleeding provoked by the intubation was also examined by another otolaryngologist 5 minutes later, who was not aware of the chosen technique to complete intubation.

Hemodynamic parameters were recorded in the operating theatre after starting standard monitoring. Measurement of hemodynamic parameters included of time interval of baseline, intubation and post-intubation 1, 3 and 5 min, respectively. Anesthesia was maintained with sevoflurane. At the end of surgery, patients were trained to breathe spontaneously. The DLT was removed when spontaneous ventilation reached a tidal volume of 8 ml/kg and the patient could respond to simple verbal commands. The patients were interviewed by an independent investigator to determine whether they were suffering from a sore throat or dysphagia the next day of post-operation. We quantified the degree of soreness of the throat and dysphagia by using a visual analogue scale ranging from 0 to 10, with VAS 0 being rated as 'none', 1-3 as 'mild', 4-6 as moderate' and 7-10 as 'severe'.

Assuming a likely difference in mean times to intubate of 10 s with a SD of 10 s, an a priori power analysis revealed a group size of n = 27 was needed to detect a difference with a power of 0.8 at α-level of 0.05. Statistical analysis was performed using the Mann-Whitney U-test for non-parametric and univariate ANOVA for parametric data. Duncan's post-hoc test was performed where appropriate. Hemodynamic data were analyzed with ANOVA for repeated measures. Data are expressed as mean (SD) where applicable or actual numbers. SPSS 16.0.1 software (Apache Software Foundation, Forest Hill, MD, USA) was used for all statistical analyses.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesiologists physical status I-III, ≧ 18 years of age, and needed double-lumen endotracheal tube (DLT) for thoracic surgery

Exclusion Criteria:

* increased risk for regurgitation and pulmonary aspiration, history of gastroesophageal reflux, and pregnancy
* a tracheostomy or prolonged ventilation on ICU was planned, patients were also excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Main outcome measure is the successful rate of the first intubation compared with the two devices | 12 month

SECONDARY OUTCOMES:
The outcome measure is the time needed to inert the DLT compared with the two devices | 12 months
The outcome measure were the hemodynamic parameters (such as mean blood pressure, and heart rate) compared with the two devices. | 12 months
The outcome measure is the incidence of complications (such as sorethroat, oral bleeding, and hypoxemia) compared with the two devices. | 12 months
  Hypoxemia is defined as the SPO2 is below 90%.

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Te Hsu, MD, Principal Investigator — Department of anesthesia, Kaoshiung medical university hospital
Locations (1):
- department of anesthesia, Kaohsiung medical university memorial hospital, Kaohsiung, Taiwan, Taiwan